CLINICAL TRIAL: NCT06558279
Title: A Randomized, Double-Blinded, Placebo-Controlled, Phase 3, Parallel-Group Design Study Evaluating the Efficacy and Safety of Efgartigimod PH20 SC Administered by Prefilled Syringe in Adult Participants With Ocular Myasthenia Gravis
Brief Title: A Study to Assess Efficacy and Safety of Efgartigimod PH20 SC in Adults With Ocular Myasthenia Gravis
Acronym: ADAPT oculus
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: argenx (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ARGX-113-2315; 2024-514133-38-00 (EU CTIS Number)
Record Dates: First submitted 2024-08-14; First posted 2024-08-16 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Myasthenia Gravis, Ocular
Keywords: Myasthenia Gravis; Ocular myasthenia
MeSH Terms: conditions — Myasthenia Gravis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Efgartigimod PH20 SC in part A+B (Experimental): Participants receiving efgartigimod PH20 SC during part A and part B
  Interventions: Combination Product: Efgartigimod PH20 SC
- Placebo PH20 SC in Part A + Efgartigimod PH20 SC in Part B (Experimental): Participants receiving placebo PH20 SC in Part A and Efgartigimod PH20 SC in Part B
  Interventions: Combination Product: Efgartigimod PH20 SC; Other: Placebo PH20 SC

INTERVENTIONS:
Combination Product: Efgartigimod PH20 SC — Subcutaneous efgartigimod PH20 SC given by prefilled syringe
Other: Placebo PH20 SC — Subcutaneous placebo PH20 SC given by prefilled syringe
  Arms: Placebo PH20 SC in Part A + Efgartigimod PH20 SC in Part B

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of efgartigimod PH20 SC given by a pre-filled syringe in adult patients with ocular myasthenia gravis. The study consists of a part A (approximately 7 weeks) and a part B (up to 2 years). In part A, half of the participants will receive efgartigimod PH20 SC and the other half will receive placebo. In part B, all participants will receive efgartigimod PH20 SC. The participants will be in the study for about up to 2 years and 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Is at least 18 years of age and the local legal age of consent for clinical studies
* Has been diagnosed with myasthenia gravis and supported by seropositivity for AChR-Ab; or abnormal neuromuscular transmission demonstrated by abnormal neurophysiology testing and history on positive edrophonium chloride testing or demonstrated improvement on MG therapy"
* Is MGFA Class I (any ocular muscle weakness)
* Has a screening and baseline MGII (PRO) ocular score of at least 6 with at least 2 ocular items with a score of at least 2

Exclusion Criteria:

* Other diseases that lead to eyelid drooping, peripheral muscle weakness, or diplopia
* Known autoimmune disease or any medical condition other than indication under study that would interfere with an accurate assessment of clinical symptoms of ocular myasthenia gravis or puts the participant at undue risk

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2024-09-18 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
MGII (PRO) ocular score change from baseline to day 29 in part A | Up to 29 days
  The Myasthenia Gravis Impairment Index (MGII) is a scoring tool measuring disease severity. It consists of 22 patient-reported outcomes (PRO) and 6 physical examinations (PE). The Ocular PRO score varies between 0 and 18. The higher the score, the more severe the disease.

SECONDARY OUTCOMES:
MGII (PRO+PE) ocular score change from baseline to day 29 in part A | Up to 29 days
  The Myasthenia Gravis Impairment Index (MGII) is a scoring tool measuring disease severity. It consists of 22 patient-reported outcomes (PRO) and 6 physical examinations (PE). The Ocular PRO score varies between 0 and 18. The ocular PE score varies between 0 and 5. The higher the score, the more severe the disease.
MG-ADL ocular domain score change from baseline to day 29 in part A | Up to 29 days
  The Myasthenia Gravis Activities of Daily Living (MG-ADL) scale assesses MG symptoms and their effects on daily activities. The ocular score varies between 0 and 16 (with 16 the most severe).
MGII total score change from baseline to day 29 in part A | Up to 29 days
  The Myasthenia Gravis Impairment Index (MGII) is a scoring tool measuring disease severity. It consists of 22 patient-reported outcomes (PRO) and 6 physical examinations (PE). The score varies between 0 and 84. The higher the score, the more severe the disease.
MGII (PE) ocular score change from baseline to day 29 in part A | Up to 29 days
  The Myasthenia Gravis Impairment Index (MGII) is a scoring tool measuring disease severity. It consists of 6 physical examinations (PE). The score varies between 0 and 5. The higher the score, the more severe the disease.
MG-ADL total score change from baseline to day 29 in part A | Up to 29 days
  The Myasthenia Gravis Activities of Daily Living (MG-ADL) scale assesses MG symptoms and their effects on daily activities. The score varies between 0 and 24 (with 24 the most severe).
MGII ocular scores changes (PRO) from baseline in part A+B | Up to 111 weeks
  The Myasthenia Gravis Impairment Index (MGII) is a scoring tool measuring disease severity. It consists of 22 patient-reported outcomes (PRO) and 6 physical examinations (PE). The Ocular PRO score varies between 0 and 18. The ocular PE score varies between 0 and 5. The higher the score, the more severe the disease.
Incidence of (serious) adverse events | Up to 111 weeks
MG-QoL15r total score changes from baseline in part A+B | Up to 111 weeks
  The Myasthenia Gravis Quality of Life 15-item scale revised (MG-QoL15r) questionnaire is a patient-reported instrument that measures the impact of MG symptoms on Quality of Life. The score varies between 0 and 30 (with 30 the lowest quality of life).
NEI VFQ-25 score changes from baseline in part A+B | Up to 111 weeks
  The 25-item National Eye Institute Visual Function Questionnaire (NEI VFQ-25) is a 25-item vision-targeted questionnaire. The score varies between 0 and 100 (with 0 being the worst score)
Percent change from baseline in total IgG levels over time in part A+B | Up to 111 weeks
Percent change from baseline in AChR-Ab levels in AChR-Ab seropositive participants over time in part A+B | Up to 111 weeks
Incidence of Anti-Drug Antibodies and Neutralizing Antibodies against efgartigimod in part A+B | Up to 111 weeks
Incidence of antibodies and Neutralizing Antibodies against rHuPH20 in part A+B | Up to 111 weeks

CONTACTS AND LOCATIONS:
Locations (102):
- United States (20):
  - HonorHealth Neurology - Bob Bové Neuroscience Institute, Scottsdale, Arizona
  - Loma Linda University Health, Loma Linda, California
  - USC Roski Eye Institute - Los Angeles, Los Angeles, California
  - University of California San Francisco, San Francisco, California
  - Neurology Offices of South Florida, Boca Raton, Florida
  - SFM Clinical Research, LLC, Boca Raton, Florida
  - Neurology Associates PA, Maitland, Florida
  - University of South Florida, Tampa, Florida
  - Northwestern Memorial Hospital, Chicago, Illinois
  - University of California Irvine, Columbia, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Duke Neurological Disorders Clinic, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Martha Morehouse Medical plaza, Columbus, Ohio
  - Penn Medicine University City, Philadelphia, Pennsylvania
  - National Neuromuscular Research Institute, Austin, Texas
  - Houston Methodist Neurological Institute, Houston, Texas
- Australia (3):
  - Box Hill Hospital, Box Hill
  - The Alfred Hospital, Melbourne
  - Gold Coast University Hospital, Southport
- Universitätsklinikum AKH Wien, Vienna, Austria
- Belgium (2):
  - UZ Leuven, Leuven
  - Hôpital de la Citadelle, Liège
- Canada (6):
  - Maritime Neurology, Halifax
  - London Health Sciences Centre, London
  - Centre Hospitalier de l'Universite de Montreal, Montreal
  - Ottawa Hospital Research Institute, Ottawa
  - Hopital de L'enfant Jesus, Québec
  - Toronto General Hospital, Toronto
- China (12):
  - Xiangya Hospital Central South University, Changsha
  - Sichuan Academy of Medical Sciences & Sichuan Provincial People's Hospital, Chengdu
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing
  - Fujian Medical University Union Hospital, Fuzhou
  - Guangdong Province Traditional Chinese Medical Hospital, Guangzhou
  - The First Affiliated Hospital of Guangzhou University Chinese Medicine, Guangzhou
  - Qilu Hospital of Shandong University, Jinan
  - The First Affiliated Hospital of Nanchang University - Xianghu Campus, Nanchang
  - Huashan Hospital Fudan University, Shanghai
  - Shijiazhuang People's Hospital - Fangbeilu Campus, Shijiazhuang
  - Tongji Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan
  - Renmin Hospital of Wuhan University - Main Campus, Wuhan
- Cyprus Institute of Neurology and Genetics, Égkomi, Cyprus
- Czechia (2):
  - Fakultni nemocnice Brno, Brno
  - Nemocnice Pardubickeho kraje, a.s., Pardubicka nemocnice, Pardubice
- Denmark (2):
  - Aarhus Universitetshospital, Aarhus N
  - Rigshospitalet, Copenhagen
- Turun Yliopistollinen Keskussairaala, Turku, Finland
- Hôpital Fondation Adolphe de Rothschild, Paris, France
- Georgia (4):
  - Petre Sarajishvili Institute of Neurology, Tbilisi
  - New Hospitals, Tbilisi
  - Pineo Medical Ecosystem, Tbilisi
  - LLC Caucasus Medical Centre, Tbilisi
- Germany (2):
  - Charité - Universitätsmedizin Berlin, Berlin
  - Universität Georg August, Göttingen
- Greece (2):
  - Eginitio Hospital, Athens
  - University General Hospital of Patras, Pátrai
- Italy (6):
  - ASST Papa Giovanni XXIII - Ospedale Papa Giovanni XXIII, Bergamo
  - IRCCS Istituto dell Scienze Neurologiche di Bologna, Bologna
  - Ospedale San Raffaele S.r.l., Milan
  - Fondazione IRCCS Istituto Neurologico Carlo Besta, Milan
  - AORN Antonio Cardarelli, Napoli
  - Azienda Ospedaliero-Universitaria Sant'Andrea, Roma
- Japan (11):
  - Chiba University Hospital, Chūōku
  - Kyushu University Hospital, Fukuoka
  - General Hanamaki Hospital, Hanamaki-shi
  - Hiroshima University Hospital, Hiroshima
  - Saitama Medical Center, Kawagoe
  - National Hospital Organization Utano National Hospital, Kyoto
  - IUHW Narita Hospital, Narita
  - National Hospital Organization Hokkaido Medical Center, Sapporo
  - Kindai University Hospital, Sayama
  - Tokyo Medical University Hospital, Shinjuku-Ku
  - Osaka University Hospital, Suita-Shi
- Leids Universitair Medisch Centrum, Leiden, Netherlands
- Poland (5):
  - MICS Centrum Medyczne Bydgoszcz, Bydgoszcz
  - Centrum Medyczne Neurologia Slaska, Katowice
  - SP ZOZ Szpital Uniwersytecki, Krakow
  - Krakowska Akademia Neurologii, Krakow
  - CLINIREM Sp z o.o., Lublin
- Portugal (2):
  - ULS de Santa Maria, EPE - Hospital de Santa Maria, Lisbon
  - ULS de Santo António, EPE - Hospital de Santo António, Porto
- Serbia (2):
  - University Clinical Center of Serbia, Belgrade
  - University Clinical Center Nis, Niš
- South Korea (3):
  - Kyungpook National University Chilgok hospital, Daegu
  - Korea University Anam Hospital, Seoul
  - Severance Hospital Yonsei University Health System, Seoul
- Spain (6):
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital del Mar, Barcelona
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario de Donostia, San Sebastián
  - Hospital Clinico Universitario de Valencia, Valencia
- Sahlgrenska Universitetssjukhuset, Gothenburg, Sweden
- Mediclinic Parkview, Dubai, United Arab Emirates
- United Kingdom (5):
  - Royal Sussex County Hospital, Brighton
  - Panthera Biopartners - Glasgow, Glasgow
  - Leeds General Infirmary, Leeds
  - Dementech Neurosciences Clinical Academic Centre, London
  - Southampton General Hospital, Southampton

IPD SHARING:
Plan to Share IPD: No